CLINICAL TRIAL: NCT03422536
Title: A Randomized, Phase II Study of Ficlatuzumab With or Without Cetuximab in Patients With Cetuximab-Resistant, Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Ficlatuzumab w/wo Cetuximab in Patients w/Cetuximab-Resistant, Recurrent or Metastatic Head/Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1710965268; NCI-2017-02209 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AV-299-17-117i (Other: Aveo Oncology and Biodesix); 1710965268 (Other: The University of Arizona Medical Center-University Campus); P30CA023074 (NIH)
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Basaloid Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Unknown Primary Origin; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IV Oropharyngeal Squamous Cell Carcinoma; Stage IVA Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVA Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVA Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IVA Oropharyngeal Squamous Cell Carcinoma; Stage IVB Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVB Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVB Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IVB Oropharyngeal Squamous Cell Carcinoma; Stage IVC Lip and Oral Cavity Squamous Cell Carcinoma; Stage IVC Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IVC Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IVC Oropharyngeal Squamous Cell Carcinoma; Head and Neck Cancer; Oropharyngeal Cancer; HNSCC; Stage IV Lip and Oral Cavity Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; Oropharyngeal Cancer; Squamous Cell Carcinoma; lip carcinoma; oral cavity carcinoma; HNSCC; Head and Neck Squamous Cell Carcinoma; AVEO
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Carcinoma, Squamous Cell; Lip Neoplasms; Mouth Neoplasms | interventions — Cetuximab; ficlatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (ficlatuzumab) (Experimental): Patients receive ficlatuzumab IV over 30-60 minutes every 2 weeks in the absence of disease progression or unaccepted toxicity. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ficlatuzumab
- Arm II (ficlatuzumab, cetuximab) (Experimental): Patients receive cetuximab IV over 60 -120 minutes and ficlatuzumab IV over 30-60 minutes every 2 weeks in the absence of disease progression or unaccepted toxicity. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: Ficlatuzumab

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm II (ficlatuzumab, cetuximab)
Drug: Ficlatuzumab — Given IV
  Other Names: Anti-HGF Monoclonal Antibody SCH900105; AV-299; SCH 900105

SUMMARY:
This randomized phase II trial studies how well ficlatuzumab with or without cetuximab works in treating patients with head and neck squamous cell carcinoma that has come back or spread to other places in the body and resistant to cetuximab treatment. Monoclonal antibodies, such as ficlatuzumab and cetuximab, may block growth signals that lets a tumor cell survive and reproduce, and helps the immune system recognize and fight head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of ficlatuzumab, with or without concurrent cetuximab, in patients with cetuximab-resistant, recurrent/metastatic head and neck squamous cell carcinoma (HNSCC) as measured by progression-free survival (PFS).

SECONDARY OBJECTIVES:

I. To describe toxicity. II. To evaluate response rate and overall survival in both treatment arms.

EXPLORATORY OBJECTIVES I. To describe patient reported quality of life

II. To evaluate the relationship between clinical outcomes (Progression-Free Survival and Response Rate) and candidate tumoral, genomic, peripheral, and immune biomarkers, potentially including but not limited to:

* Tumor Hepatocyte Growth Factor (HGF) and tyrosine-protein kinase Met (cMet) expression
* mutations in PIK3CA, phosphatase and tensin homolog (PTEN), and HumanRAS proto-oncogene (HRAS);
* peripheral serum biomarkers including HGF, soluble HGF, and interleukin 6 (IL6);
* peripheral lymphocyte populations;
* archived and baseline immune infiltrate;
* tumor Human Papilloma Virus (HPV) status.

OUTLINE: Patients are randomized into 1 of 2 arms.

Arm I: Patients receive ficlatuzumab intravenously (IV) over 30-60 minutes every 2 weeks in the absence of disease progression or unaccepted toxicity. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Arm II: Patients receive cetuximab IV over 60 -120 minutes and ficlatuzumab IV over 30-60 minutes every 2 weeks in the absence of disease progression or unaccepted toxicity. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

- Patients must have histologically confirmed HNSCC from any primary site, except nasopharyngeal if World Health Organization (WHO) Type III (non-keratinizing and Epstein-Barr virus (EBV)-positive)).

Eligible histologies include:

* Basaloid, poorly differentiated, and undifferentiated carcinoma histologies.
* Nasopharyngeal carcinoma, WHO Type I and II (keratinizing, non-EBV positive).
* Paranasal sinus, lip and external auditory canal sites.
* Squamous cell carcinoma of unknown primary, clearly related to the head and neck.

Note: Documentation of primary site diagnosis must be submitted with the registration request.

* Patients must have recurrent and/or metastatic disease, fulfilling at least one of the criteria defined below:
* Incurable disease as assessed by surgical or radiation oncology;
* Metastatic (M1) disease;
* Persistent or progressive disease following curative-intent radiation, and not a candidate for surgical salvage due to incurability or morbidity. Note: Patients who decline radical surgery are eligible.
* For patients with oropharyngeal primary site or unknown primary site only: Patients must have known tumoral HPV status (p16). (Acceptable standards include p16 immunohistochemistry (where a tumor is classified as p16-positive when showing diffuse nuclear and cytoplasmic staining in at least 70% of tumor cells) and/or assessment of HPV DNA.) Note: For these subjects, documentation of p16 status must be submitted with the registration packet.
* Patients must be cetuximab-resistant by fulfilling at least one of the two criteria defined below:
* Disease persistence or recurrence within 6 months of completing definitive radiotherapy with concurrent cetuximab for locally advanced disease. Induction chemotherapy, if given, may or may not have included cetuximab.
* Disease progression during, or within 6 months, of cetuximab treatment in the recurrent and/or metastatic setting.

Note: Prior cetuximab exposure may have occurred in any line of therapy (first line, second line, etc.) and is not required to be the most recent therapy received.

* Patients must be platinum-resistant or platinum-ineligible by fulfilling at least one of the three criteria defined below:
* Disease persistence or recurrence within 6 months of completing definitive radiotherapy for locally advanced disease, where platinum chemotherapy was administered as a component of induction and/or concurrent systemic treatment.
* Disease progression during, or within 6 months, of treatment with platinum chemotherapy (e.g., carboplatin or cisplatin) in the recurrent and/or metastatic setting.
* The patient is not an acceptable candidate for platinum chemotherapy due to medical comorbidities, in the judgment of the local investigator.

Note: Prior platinum exposure may have occurred in any line of therapy (first line, second line, etc.) and is not required to be the most recent therapy received.

- Patients must have prior exposure to an anti-PD1 (programmed cell death protein 1) or anti-PDL1 (programmed cell death ligand 1) monoclonal antibody (mAb), if eligible for immunotherapy in the judgment of the local investigator.

Note: Prior exposure to investigational immunotherapies, including anti-CTLA4 (cytotoxic T-lymphocyte-associated antigen 4), anti-OX40, anti-CD40 (cluster of differentiation 40), anti-CD27, anti-TNFR (tumor necrosis factor receptor) antibodies or other investigational immunotherapies, is acceptable.

* Patients must have Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 at time of informed consent (see Appendix B).
* Patients must be age ≥ 18 years.
* Patients must consent to a research biopsy of tumor tissue at baseline, for conduct of correlative studies. In cases where a fresh biopsy is not feasible (i.e., if an accessible tumor site cannot be biopsied with acceptable clinical risk), archival tissue may be submitted instead, after discussion with and approval by the Sponsor-Investigator.
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1 (see section 6) per scan within 28 days prior to registration.
* Patients must have adequate electrolytes, liver, renal, and hematology function as defined below within 28 days of registration:
* Absolute neutrophil count (ANC) ≥ 1500/mm3
* Platelet count (PLT) ≥ 75,000/mm3
* Creatinine clearance ≥ 30 mL/min per estimated by the Cockraft-Gault formula:
* Calculated Creatinine Clearance = [(140-age) X (actual body weight in kg) X (0.85 if female)]/(72 X serum creatinine)

  * Total bilirubin ≤ 1.5 times upper-limit of normal (ULN)
* AST (aspartate aminotransferase) ≤ 3 times ULN
* ALT (alanine aminotransferase) ≤ 3 times ULN
* Magnesium ≥ 1.2 mg/dL or 0.5 mmol/L
* Corrected Calcium ≥ 8.0 mg/dL or 2.0 mmol/L
* Potassium ≥ 3.0 mmol/L (Note: Patients may be supplemented to achieve acceptable electrolyte values.)
* Serum albumin ≥ 25 g/L (≥ 2.5 g/dL)
* Patients must sign written informed consent prior to beginning study screening procedures. Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Women of child-bearing potential (WOCBP) must agree to have a pregnancy test within 14 days prior to registration and a repeated test within 3 days of the first dose of ficlatuzumab.
* Patients must agree to use highly effective contraceptive measures while on study and for 60 days after the last dose of study drug. This includes: Men of reproductive potential AND women of childbearing potential.
* Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm).

Exclusion Criteria

* Nasopharyngeal primary site if WHO Type III (non-keratinizing and EBV-positive as established at the local site).
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent.
* Prior treatment with an HGF/cMet inhibitor such as rilotumumab, crizotinib, MetMAb, or tivantinib (ARQ197).
* Uncontrolled central nervous system (CNS) metastases, including leptomeningeal metastases, are not allowed.

Note: Subjects with previously treated brain metastases will be allowed if the brain metastases have been stable without steroid treatment for at least 2 weeks (radiotherapy or surgery).

* Failure to recover to Grade 1 or baseline from all toxic effects of previous chemotherapy, radiation therapy, biologic therapy, immunotherapy, and/or experimental therapy, with the exception of:
* Alopecia,
* Grade ≤ 2 peripheral neuropathy,
* Grade ≤ 2 cetuximab-related rash or other skin changes,
* Hypomagnesemia (acceptable values detailed in the exclusion criteria below),
* Hypokalemia (acceptable values detailed in the exclusion criteria below), and
* The acceptable ANC and PLT inclusion criteria values above.
* Treatment with cetuximab 2 weeks prior to the first dose of study drug. A washout period of 2 weeks from prior cetuximab is required if applicable.
* Treatment with cytotoxic chemotherapy, targeted therapy, immunotherapy or investigational drug 3 weeks prior to the first dose of study drug. A washout period of 3 weeks from any prior cytotoxic chemotherapy, targeted therapy, immunotherapy or investigational drug is required, if applicable.
* Significant underlying pulmonary disease, including pulmonary hypertension or interstitial pneumonitis.
* Peripheral edema ≥ Grade 2 per NCI-CTCAE version 4.0.
* Significant cardiovascular disease, including:
* Cardiac failure New York Heart Association (NYHA) class III or IV.
* Myocardial infarction within 6 months prior to registration.
* Severe or unstable angina within 6 months prior to registration.
* History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation).
* Cardiac arrhythmia requiring anti-arrhythmic medication(s). (Beta-blockers, calcium channel blockers, and digoxin administered for the purpose of rate control of supraventricular tachycardia, including atrial fibrillation and atrial flutter, are not classified as anti-arrhythmic medications for purposes of trial eligibility.)
* Significant thrombotic or embolic events within 28 days prior to registration. (Significant thrombotic or embolic events include but are not limited to stroke or transient ischemic attack (TIA). Catheter-related thrombosis is not a cause for exclusion. Diagnosis of deep vein thrombosis or pulmonary embolism is allowed if it occurred > 28 days prior to registration and the patient is asymptomatic and stable on anti-coagulation therapy.)
* Any other medical condition (e.g., alcohol abuse) or psychiatric condition that, in the opinion of the local Investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.
* History of second malignancy within 2 years prior to registration except:
* Excised and cured non-melanoma skin cancer,
* Carcinoma in situ of breast or cervix,
* Superficial bladder cancer,
* Stage I differentiated thyroid cancer that is resected or observed,
* pT1a /pT1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection, or

  * cT1a/cT1b prostate cancer treated with brachytherapy or external beam radiation therapy with normal PSA since radiation.
* Not completely recovered from any previous surgery. Note: Complete recovery is in the opinion of the treating investigator. Consult the Sponsor-Investigator, if needed.
* Active systemic infection requiring systemic antibiotics or antifungals within 7 days prior to first dose of study drug, except tetracycline family antibiotics (tetracycline, doxycycline, minocycline) administered for the management of cetuximab-related rash may be continued per the Investigator's judgment.

Note: Active topical infections (for example oral thrush) do not exclude a subject even if treated with systemic antibiotics or systemic antifungals.

* History of severe infusion reaction to cetuximab or a monoclonal antibody.
* Known to be Human immunodeficiency virus (HIV) positive. Note: HIV testing is not required for entry into this protocol.
* Women who are pregnant or breastfeeding. (A negative urine pregnancy test must be confirmed within 14 days of registration and repeated within 3 days of the first dose of study drug.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie E. Bauman, MD, MPH, Principal Investigator — The University of Arizona
Locations (6):
- United States (6):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Bauman JE, Saba NF, Roe D, Bauman JR, Kaczmar J, Bhatia A, Muzaffar J, Julian R, Wang S, Bearelly S, Baker A, Steuer C, Giri A, Burtness B, Centuori S, Caulin C, Klein R, Saboda K, Obara S, Chung CH. Randomized Phase II Trial of Ficlatuzumab With or Without Cetuximab in Pan-Refractory, Recurrent/Metastatic Head and Neck Cancer. J Clin Oncol. 2023 Aug 1;41(22):3851-3862. doi: 10.1200/JCO.22.01994. Epub 2023 Mar 28. PMID 36977289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted at the University of Arizona, Emory University, Fox Chase Cancer Center, Medical University of South Carolina, Yale Cancer Center, and Moffitt Cancer Center. The study opened to accrual on 12/05/2017 and closed to accrual on 12/05/2020. Potential patients were identified in the cancer center clinic by study investigators or referred. Weekly tumor board meetings are held at each institution where patients are discussed and referred to clinical trials.
Pre-assignment Details: Of the 78 patients who signed consent, only 60 were randomized. 18 patients were excluded, 15 were determined to be ineligible after the screening period and 3 declined to participate after signing consent.
Period: Randomized
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab)
Started | 27 | 33
Completed | 26 | 32
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 1
Period: Allocation - Received Intervention
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab)
Started | 26 | 32
Completed | 0 | 1
Not Completed | 26 | 31
Not completed — Disease progression | 19 | 25
Not completed — Death | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab) | Total
Number analyzed (Participants) | 27 | 33 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [55 to 70] | 63 [59 to 71] | 63.5 [56.75 to 70.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 21 | 30 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 23 | 29 | 52
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 24 | 30 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 33 | 60
Primary Site [Number; unit: participants]
  Oral Cavity | 8 | 6 | 14
  Oropharynx | 11 | 20 | 31
  Larynx | 3 | 4 | 7
  Nasopharynx | 2 | 1 | 3
  Paranasal sinus | 2 | 0 | 2
  External auditory canal | 0 | 1 | 1
  Unknown primary | 1 | 1 | 2
HPV status [Number; unit: participants]
  Positive | 11 | 17 | 28
  Negative | 16 | 16 | 32
Median months since last cetuximab treatment [Median (Inter-Quartile Range); unit: Months] | 2.7 [0.9 to 13.1] | 3.6 [1.4 to 9.3] | 3.5 [1.1 to 9.7]
History of platinum [Number; unit: participants] | 27 | 32 | 59
History of anti-PD-1 (checkpoint protein) monoclonal antibody (mAb) treatment [Number; unit: participants] | 25 | 31 | 56
Eastern Cooperative Oncology Group Performance Status (ECOG- PS) [Number; unit: participants]
  Asymptomatic (0) - Fully active, able to carry on all pre-disease performance without restriction | 9 | 6 | 15
  Symptomatic (1) - restricted in physically strenuous activity but able to carry out light work | 18 | 27 | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Will be estimated for each arm using a Kaplan-Meier curve.
Time Frame: From the date of randomization until the date of progression or death, assessed up to 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab)
Number analyzed (Participants) | 26 | 32
months | 1.8 [1.7 to NA] — The Upper Confidence Interval was not computable as 50% of the group had not reached median PFS. | 3.7 [2.3 to NA] — The Upper Confidence Interval was not computable as 50% of the group had not reached median PFS.
Statistical Analysis 1: Comparison: Arm II (Ficlatuzumab, Cetuximab); Test type: Equivalence — The pre-specified significance criteria were met by exclusion of the historical control PFS of 2.0 months. As confirmation, the one-sample log rank test was computed with expected survival estimated using an exponential distribution of 2.0 months; p = .04, Log Rank — The a priori threshold for statistical significance is <.05

2. Secondary Outcome: Percentage of Participants With Dose Limiting Toxicities or Adverse Events
Description: The percentage of participants with dose limiting toxicities in each dosing cohort will be reported, as will the percentage of participants with adverse events in accordance with National Cancer Institute Common Terminology Criteria for Adverse Events version 4 grading criteria. Will be tabulated and reported with 95% exact confidence intervals.
Time Frame: Up to 2 years
Population: The most common AEs are notated below.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab)
Number analyzed (Participants) | 26 | 32
percentage of participants
  hypoalbuminemia | 66 | 76
  Edema | 25 | 44
  Acneiform rash | 12 | 82
  Pneumonitis | 8 | 3

3. Secondary Outcome: Overall Survival (OS)
Description: Will be estimated for each arm using a Kaplan-Meier curve.
Time Frame: From the date of randomization until the date of death, assessed up to 2 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab)
Number analyzed (Participants) | 26 | 32
months | 6.4 [3.0 to NA] — Note: The upper confidence interval for the Median Overall Survival was not computable as 50% of the group did not reach median OS | 7.4 [4.7 to NA] — Note: The upper confidence interval for the Median Overall Survival was not computable as 50% of the group did not reach median OS

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST v1.1) for target lesions and assessed by CT/MRI w/ contrast: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), the regression of all Target lesions (the sum) by 30% with no progression of Non-targets or presence of new lesion; Overall Response (OR) = CR + PR. Will be tabulated and reported with 95% exact confidence intervals.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab)
Number analyzed (Participants) | 26 | 32
Participants | 1 | 6

5. Other Pre Specified Outcome: Change in Quality of Life
Description: Will be assessed by Foundation for the Accreditation of Cellular Therapy Head and Neck Questionnaire.
Time Frame: Pre-study (within 4 weeks of study registration) and Week 4, Cycle 2 of Intervention
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Tumor Biomarker Analysis
Description: Will evaluate the relationship between clinical outcomes (progression free survival, response rate) and candidate tumoral biomarkers: Tumor HGF and cMET expression. The relationship with clinical response will be assessed.
Time Frame: Up to 2 years
Population: Exploratory biomarker analysis was only conducted for the combination arm. The monotherapy arm closed for futility. It would be costly and would not add value to study biomarkers in the setting of an inactive agent to perform analyses for the monotherapy arm thus the limited funds available for correlatives were allocated to the combination arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab)
Number analyzed (Participants) | 0 | 26
Participants
  HPV-negative patients |  | 13
  HPV-positive patients |  | 13
  HGF - HPV-positive |  | 13
  HGF - HPV-negative |  | 13
  C-met positive in HPV-negative patients: number analyzed (Participants) | 0 | 13
  C-met positive in HPV-negative patients |  | 9
  C-met positive in HPV-positive patients: number analyzed (Participants) | 0 | 13
  C-met positive in HPV-positive patients |  | 2
Statistical Analysis 1: Comparison: Arm II (Ficlatuzumab, Cetuximab); c-Met positivity was compared across groups: HPV+ vs HPV-; Test type: Superiority; p = .005, Regression, Cox
Statistical Analysis 2: Comparison: Arm II (Ficlatuzumab, Cetuximab); Post-hoc comparison of progression free survival (PFS) in cMet positive vs. c-Met negative patients; Test type: Superiority; p = .02, Log Rank; Cox Proportional Hazard = 0.3, 95% CI 2-sided [0.1 to 0.8]
Statistical Analysis 3: Comparison: Arm II (Ficlatuzumab, Cetuximab); Post hoc comparison of PFS in the combination arm by HPV subgroup, adjusted for prognostic factors marginally associated with HPV status (P , .10), was assessed using Cox proportional hazards models. Here we are looking at cMet positivity in HPV- patients in the combination arm; Test type: Superiority; p = 0.03, Log Rank; Cox Proportional Hazard = 0.1, 95% CI 2-sided [0.03 to 0.8]
Statistical Analysis 4: Comparison: Arm II (Ficlatuzumab, Cetuximab); Post hoc comparison of PFS in the combination arm by HPV subgroup, adjusted for prognostic factors marginally associated with HPV status (P , .10), was assessed using Cox proportional hazards models. Here we are looking at cMet positivity in HPV+ patients in the combination arm; Test type: Superiority; p = .20, Log Rank; Cox Proportional Hazard = 3.2, 95% CI 2-sided [0.6 to 17.5]
Statistical Analysis 5: Comparison: Arm II (Ficlatuzumab, Cetuximab); Post-hoc comparison of progression free survival (PFS) in HGF positive vs. HGF negative patients; Test type: Superiority; p = .10, Log Rank; Cox Proportional Hazard = 1.4, 95% CI 2-sided [0.9 to 2.0]
Statistical Analysis 6: Comparison: Arm II (Ficlatuzumab, Cetuximab); Post hoc comparison of PFS in the combination arm by HPV subgroup, adjusted for prognostic factors marginally associated with HPV status (P , .10), was assessed using Cox proportional hazards models. Here we are looking at HGF expression in HPV- patients in the combination arm; Test type: Superiority; p = .60, Log Rank; Cox Proportional Hazard = 1.4, 95% CI 2-sided [0.4 to 4.7]
Statistical Analysis 7: Comparison: Arm II (Ficlatuzumab, Cetuximab); Post hoc comparison of PFS in the combination arm by HPV subgroup, adjusted for prognostic factors marginally associated with HPV status (P < .10), was assessed using Cox proportional hazards models. Here we are looking at HGF expression in HPV+ patients in the combination arm; Test type: Superiority; p = .07, Log Rank; Cox Proportional Hazard = 3.4, 95% CI 2-sided [0.9 to 13.1]

7. Other Pre Specified Outcome: Genomic Biomarker Analysis
Description: To evaluate the relationship between clinical outcomes (Progression-Free Survival and Response Rate) and candidate genomic biomarkers: mutations in PIK3CA, PTEN, and HRAS
Time Frame: Up to 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Peripheral Biomarker Analysis
Description: Will evaluate the relationship between clinical outcomes (progression free survival, response rate) and candidate peripheral biomarkers: peripheral serum biomarkers including HGF, soluble HGF, and IL6; peripheral lymphocyte populations. The relationship with clinical response will be assessed.
Time Frame: Up to 2 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Immune Biomarker Analysis
Description: Will evaluate the relationship between clinical outcomes (progression free survival, response rate) and candidate immune biomarkers: archived and baseline immune filtrate; tumor HPV status. The relationship with clinical response will be assessed.
Time Frame: Up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected staring at Cycle1 Day1 and continued at each study visit during the treatment phase. I.e., day 1 and day 15 of each 28-day cycle, and any unplanned visits. Subjects are followed for AEs for at least 60 days after the last dose of study drug(s) or until the initiation of subsequent antineoplastic therapy, whichever is earlier, up to 2 years. During the 60-day follow up, AEs are assessed at each scheduled follow-up visit, and any unplanned contacts.
Description: Only AEs meeting one of the below criteria were collected:
  * Any AE that is Grade 3 or >
  * Any AE that results in submission of a serious adverse event(SAE)
  * Any intolerable Grade 2 AE
  * Any Grade AE resulting in a dose reduction of study drugs
  * Any Grade 2 laboratory or vital sign values that are deemed clinically significant by the treating investigator
  * Any Grade AE in the following categories:
    * Rash
    * Diarrhea
    * Edema, peripheral
    * Edema, head, face and neck
    * Hypoalbuminemia
Arm/Group | Arm I (Ficlatuzumab) | Arm II (Ficlatuzumab, Cetuximab)
All-Cause Mortality (participants affected / at risk) | 1/26 | 3/32
Serious Adverse Events (participants affected / at risk) | 7/26 | 18/32
Other Adverse Events (participants affected / at risk) | 24/26 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Ficlatuzumab) (N=26) | Arm II (Ficlatuzumab, Cetuximab) (N=32)
Pharyngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Facial edema (General disorders) | 1 (1) | 0 (0)
Limb edema (General disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2)
Oral Cavity Hemmorhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin and soft tissue infection (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 4 (4)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Genitourinary infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mitral Regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Ficlatuzumab) (N=26) | Arm II (Ficlatuzumab, Cetuximab) (N=32)
Oral infection (Infections and infestations) | 3 (3) | 2 (2)
Facial Edema (General disorders) | 5 (5) | 4 (4)
Edema limbs (General disorders) | 10 (10) | 14 (14)
Hypoalbumenia (Metabolism and nutrition disorders) | 17 (17) | 24 (24)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (4)
Rash: Maculopapular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (14)
Rash: acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 26 (26)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 2 (2)
Bacteremia (Infections and infestations) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 6 (6)
Genitourinary infection (Infections and infestations) | 0 (0) | 3 (3)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Increased AST and/or ALT (Investigations) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Weight loss (Investigations) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Oral mucositis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03422536/Prot_SAP_003.pdf
  • Informed Consent Form (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT03422536/ICF_001.pdf